CLINICAL TRIAL: NCT02400086
Title: Study of Bacterial Colonization of the Respiratory Tract in Long-term Tracheostomized Patients With Neurological or Neuromuscular Disease
Brief Title: Bacterial Colonization in Tracheostomized Patients With Neurological or Neuromuscular Disease
Acronym: ECOTRACH
Status: Completed | Type: Observational
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Sponsor
Other Study IDs: 15004
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Infectious Disorder of Trachea; Respiratory Tract Infections; Mechanical Ventilation Complication
Keywords: neuroligical or neuromuscular diseases; bacterial respiratory tract flora; long term tracheostomy
MeSH Terms: conditions — Respiratory Tract Infections; Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients with neurological or neuromuscular diseases may need a long-term tracheostomy to improve their respiratory function. Bacterial flora and bacterial drug resistance in the respiratory tract have never been studied until then for this type of patient in spite of their frequent hospital stay, their regular exposition to antibiotics and their susceptibility to swallowing disorders due to their pathology. This study is based on a single tracheal aspirate within the 48 first hours of the patient stay for a ventilation check up beside any infectious context to describe the basal bacterial respiratory flora.

DETAILED DESCRIPTION:
At their admission in Raymond Poincaré hospital in the long-term ventilation unit for a ventilation check-up, patients with a long-term tracheostomy and suffering from a neurological or neuromuscular disease will be included in the study if they have no sign of pneumonia and no contact with a hospital structure within a month. These exclusion criteria allow to focus on non-decompensating patient with a respiratory flora not hospital-acquired and not modified by antibiotics.

The doctor in charge of the patient will fill a questionnaire with the help of the patients or the patient's family with several items as date of tracheostomy, history of respiratory infections, history of hospitalization, characteristics of ventilation (presence of a cannula, frequency of change of filter, type of water use in the humidifier…). Beside, a tracheal aspirate will be collected and send to the microbiology laboratory for bacterial culture. The tracheal aspirate will be supported as a usual clinical tracheal aspirate but each bacterial specie will be quantify and identify by mass spectrometry. Antimicrobial susceptibility testing will be performed only for potential pathogenic species with a cut-off at 105.

ELIGIBILITY:
Inclusion Criteria:

* Patient of majority age who signed the information note
* Tracheostomized patient for more than 6 months for a neurological or neuromuscular disease leaving in the community and hospitalized in Raymond Poincaré hospital for less than 48 hours

Exclusion Criteria:

* Refusal to take part of the study
* Not membership in a national insurance scheme
* Patient under guardianship or curatorship
* More than 48 hours hospitalization before tracheal aspirate
* Hospitalization in the previous month
* Evolutionary pneumonia at the admission or in the previous month (fever >38.4°C with respiratory signs of pneumonia as cough, increase of the dyspnea, increase of expectorations associated with radiological opacities of recent appearance)
* Non-chronical antibiotic treatment in the previous month
* Patient already included during a previous hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with a long-term tracheostomy and suffering from a neurological or neuromuscular disease
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2015-02; Primary Completion 2017-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Description of the bacterial flora of the respiratory tract identify by tracheal aspirate at the hospital admission of long-term tracheostomized patients | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Margaux Lepainteur, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Raymond Poincaré, Garches, France